CLINICAL TRIAL: NCT05844592
Title: A First-in-Human, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of INV-101 Administered Orally to Healthy Adult Subjects
Brief Title: First in Human, Single Ascending Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: INV101-01
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- A (Placebo Comparator): Dose A
  Interventions: Drug: INV-101
- B (Placebo Comparator): Dose B
  Interventions: Drug: INV-101
- C (Placebo Comparator): Dose C
  Interventions: Drug: INV-101
- D (Placebo Comparator): Dose D
  Interventions: Drug: INV-101
- E (Placebo Comparator): Dose E
  Interventions: Drug: INV-101

INTERVENTIONS:
Drug: INV-101 — subjects will be randomized 3:1 ratio

SUMMARY:
The goal of this study is to evaluate the safety and tolerability of single ascending oral doses of INV-101 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female (of non-childbearing potential only), 19-55 years of age, inclusive, at the screening visit.
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at the screening visit.

Exclusion Criteria:

* Mentally or legally incapacitated or had significant emotional problems at the time of the screening visit or expected during the conduct of the study.
* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-07-16 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
AE | 2 weeks
  Number and severity of treatment-emergent adverse events (TEAEs) following single oral doses of INV-101 and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Minjeong Kim, Master, Study Director — New Drug development Center
Locations (1):
- Innovo Therapeutics, Inc., Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No